CLINICAL TRIAL: NCT05638737
Title: A Phase IIa, Randomized, Double-blind, Placebo-controlled Study to Evaluate Safety, Tolerability, and Pharmacodynamics of AZD4831 (Mitiperstat) in Participants With Non-cirrhotic Non-alcoholic Steatohepatitis (NASH) With Fibrosis
Brief Title: A Study in Participants With Non-cirrhotic NASH With Fibrosis
Acronym: COSMOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D6581C00001
Record Dates: First submitted 2022-10-03; First posted 2022-12-06 (Actual); Results first posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Non-Cirrhotic Non-alcoholic Steatohepatitis With Fibrosis
Keywords: NASH; Non-Cirrhotic; Steatohepatitis
MeSH Terms: conditions — Fatty Liver | interventions — AZD4831

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AZD4831 (Experimental): AZD4831
  Interventions: Drug: AZD4831
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AZD4831 — AZD4831
  Arms: AZD4831
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-group, multicenter trial. Participants will be in the trial for up to 24 weeks, including a screening period lasting up to 8 weeks, a 12-week treatment period, and a 4-week safety follow-up period

Participants are not expected to directly benefit from treatment during this trial. Participants will help researchers learn more about and how to develop AZD4831 to treat NASH.

DETAILED DESCRIPTION:
A randomized, double blind, placebo-controlled, parallel-group, multicenter study including a maximum of approximately 90 randomized adult participants with biopsy-proven non-cirrhotic non-alcoholic steatohepatitis (NASH) with fibrosis (NAS ≥ 4, fibrosis stages F1, F2, F3). The study will be conducted at approximately 48 sites across approximately 9 countries.

During screening, the participants will be checked for eligibility and enrolled in the study. Following a 8-week screening period, approximately 90 participants will be randomized in a 1:1 ratio to once daily dosing of AZD4831 or placebo. All participants will be treated once daily with AZD4831 or placebo for 12 weeks. The safety, tolerability, and pharmacodynamics will be evaluated at 12 weeks. This is the first clinical study to test AZD4831 in participants with non-cirrhotic NASH with fibrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be ≥ 18 to ≤ 75 years of age at the time of signing the informed consent.
2. Histological confirmed NASH per Clinical Research Network (CRN) criteria as diagnosed by liver biopsy (within 12 months prior screening, participants without historical biopsy should be willing to undergo a liver biopsy at screening) fulfilling all of the following criteria:

   * NAS ≥ 4 with a score of ≥ 1 for each component: steatosis, lobular inflammation and ballooning
   * Presence of fibrosis F1, F2-F3
3. One increased serum ALT measurement (ALT > ULN) at screening, and historical local serum ALT level (> ULN [41 U/L for men and 31 U/L for women] but < 300 U/L) on ≥ 1 occasion in the 6 months prior to screening.

Exclusion Criteria:

1. Liver disease of other etiologies (eg, alcoholic steatohepatitis; drug-induced, viral, or autoimmune hepatitis; primary biliary cirrhosis; primary sclerosing cholangitis; hemochromatosis; alpha 1 antitrypsin deficiency; Wilson's disease).
2. History of excessive alcohol consumption, defined as an average weekly intake of > 21 drinks/week for males or > 14 drinks/week for females. One drink is equivalent to 14 g alcohol.
3. Recent (within 3 months of randomization) use of drugs approved for weight loss (eg, orlistat, bupropion/naltrexone, phentermine-topiramate, phentermine, lorcaserin), as well as those drugs used off-label.
4. High dose vitamin E (> 400 IU) unless on a stable dose within 6 months of screening.
5. Recent (within 6 months of screening) use of therapies associated with development of NAFLD (eg, systemic corticosteroids, methotrexate, tamoxifen, amiodarone, or long-term use of tetracyclines).
6. Recent (within 6 months of screening) use of obeticholic acid or other therapy under investigation for NASH.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (54):
- United States (16):
  - Research Site, Chandler, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Chula Vista, California
  - Research Site, Montclair, California
  - Research Site, Orange, California
  - Research Site, Redondo Beach, California
  - Research Site, Stanford, California
  - Research Site, Jacksonville, Florida
  - Research Site, Lakeland, Florida
  - Research Site, Miami, Florida
  - Research Site, Las Vegas, Nevada
  - Research Site, Yonkers, New York
  - Research Site, Morehead City, North Carolina
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
- Argentina (5):
  - Research Site, CABA
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Mar del Plata
  - Research Site, Pilar
  - Research Site, Ramos Mejía
- Denmark (5):
  - Research Site, Aarhus N
  - Research Site, Esbjerg
  - Research Site, København NV
  - Research Site, København Ø
  - Research Site, Køge
- Italy (7):
  - Research Site, Catania
  - Research Site, Foggia
  - Research Site, Milan
  - Research Site, Roma
  - Research Site, Rozzano
  - Research Site, San Giovanni Rotondo
  - Research Site, Torino
- Mexico (6):
  - Research Site, Boca del Rio
  - Research Site, Cuauhtémoc
  - Research Site, Guadalajara
  - Research Site, Mexico City
  - Research Site, México
  - Research Site, Monterrey
- Norway (5):
  - Research Site, Gjøvik
  - Research Site, Grålum
  - Research Site, Lørenskog
  - Research Site, Oslo
  - Research Site, Tromsø
- Research Site, Lisbon, Portugal
- Spain (7):
  - Research Site, A Coruña
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Pozuelo de Alarcón
  - Research Site, Santander
  - Research Site, Valencia
- Sweden (2):
  - Research Site, Linköping
  - Research Site, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Armisen J, Flor A, Eriksson J, Nelander K, Bhattacharya CS, Sunnaker M, Carter D, Trebski M, Gardmark E, Aurell M, Whatling C, Challis B, Vespasiani-Gentilucci U; COSMOS Investigators. A Phase 2a Trial of Myeloperoxidase Inhibitor Mitiperstat in Non-Cirrhotic Metabolic Dysfunction-Associated Steatohepatitis. Liver Int. 2025 Nov;45(11):e70406. doi: 10.1111/liv.70406. PMID 41108609
- See also: D6581C00001-Redacted_SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6581C00001&attachmentIdentifier=f4f4aafa-cde4-46ed-bc5d-2b203ca6c82c&fileName=D6581C00001-Redacted_SAP.pdf&versionIdentifier=
- See also: D6581C00001_Redacted_CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6581C00001&attachmentIdentifier=15ec95e6-9a84-4ee3-bcd8-7b9c10d57907&fileName=D6581C00001_Redacted_CSP.pdf&versionIdentifier=
- See also: d6581C00001-Redacted_CSR_Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6581C00001&attachmentIdentifier=de017700-4bcb-497c-995e-0b09e6f3cec6&fileName=d6581C00001-Redacted_CSR_Synopsis.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Once-daily dosing of Placebo for 12 weeks
- Treatment: Once-daily dosing of 5mg mitiperstat for 12 weeks
Period: Overall Study
Arm/Group | Placebo | Treatment
Started | 56 | 56
Completed | 52 | 49
Not Completed | 4 | 7
Not completed — Withdrawal by Subject | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Placebo | Total
Number analyzed (Participants) | 56 | 56 | 112
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52 (13.1) | 53.7 (9.7) | 52.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 27 | 49
  Male | 34 | 29 | 63
Race/Ethnicity, Customized [Number; unit: Participants]
  HISPANIC OR LATINO | 29 | 29 | 58
  NOT HISPANIC OR LATINO | 27 | 27 | 54
Race/Ethnicity, Customized [Number; unit: Participants]
  AMERICAN INDIAN OR ALASKA NATIVE | 0 | 0 | 0
  ASIAN | 1 | 2 | 3
  BLACK OR AFRICAN AMERICAN | 0 | 0 | 0
  MULTIPLE | 1 | 0 | 1
  NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | 0 | 0 | 0
  NOT REPORTED | 2 | 0 | 2
  OTHER | 6 | 4 | 10
  WHITE | 46 | 50 | 96

OUTCOME MEASURES:

1. Primary Outcome: Relative to Baseline Alanine Aminotransferase (ALT)
Description: ALT at 12 weeks relative to baseline. ALT is measured in Units per litre (U/L)
Time Frame: Measurements on Baseline, Week 2, Week 4, Week 8, Week 12 and Week 16. Change reported from Baseline to Week 12.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Ratio
Groups:
- Mitiperstat (5mg): Once-daily dosing of 5mg mitiperstat for 12 weeks
Arm/Group | Mitiperstat (5mg) | Placebo
Number analyzed (Participants) | 56 | 56
Ratio | 0.959 [0.885 to 1.040] | 0.895 [0.824 to 0.972]
Statistical Analysis 1: Comparison: Mitiperstat (5mg) vs Placebo; Test type: Superiority — One-sided test where a negative change in relative to baseline is favourable; p = 0.893, Mixed Models Analysis; Participant as random effect; treatment, visit and trt:vis interaction as fixed effects; baseline ALT as covariate. Model uses log-scaled variables; %-change in relative to base vs placebo = 7.5, 95% CI 2-sided [-4.1 to 20.5]

2. Secondary Outcome: Relative to Baseline Pro-C3
Description: Pro-C3 at 12 weeks relative to baseline. Pro-C3 is measured in nanograms per milliliter (ng/mL).
Time Frame: Measurements on Baseline, Week 4 and Week 12
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Mitiperstat (5mg) | Placebo
Number analyzed (Participants) | 56 | 56
Ratio | 1.009 [0.960 to 1.060] | 1.018 [0.971 to 1.068]
Statistical Analysis 1: Comparison: Mitiperstat (5mg) vs Placebo; Test type: Superiority — One-sided test where a negative change in relative to baseline is favourable; p = 0.396, Mixed Models Analysis; Participant as random effect; treatment, visit and trt:vis interaction as fixed effects; baseline Pro-C3 as covariate. Model uses log-scaled variables; %-change in relative to base vs placebo = -0.9, 95% CI 2-sided [-7.5 to 6.1]

ADVERSE EVENTS:
Time Frame: Adverse events was collected from time of first dose throughout the treatment period and including the follow-up period, a planned period of 16 weeks. The only exception is related to the predose orthostatic test at Visit 4: If orthostatic hypotension was confirmed, it would be reported as an AE, and symptoms related to the measurement of orthostatic vitals if present should also be reported as an AE.
Arm/Group | Treatment | Placebo
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/56 | 3/56
Other Adverse Events (participants affected / at risk) | 33/56 | 36/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=56) | Placebo (N=56)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=56) | Placebo (N=56)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Faeces hard (Gastrointestinal disorders) | 0 (0) | 2 (2)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Illness (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Hepatitis alcoholic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergy to arthropod bite (Immune system disorders) | 1 (1) | 0 (0)
Food allergy (Immune system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 2 (2) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypovitaminosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (3) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (5)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Anal pruritus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-03-20): https://cdn.clinicaltrials.gov/large-docs/37/NCT05638737/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-29): https://cdn.clinicaltrials.gov/large-docs/37/NCT05638737/SAP_001.pdf